CLINICAL TRIAL: NCT07275060
Title: Immunogenicity and Safety of 2 Doses of Avian Influenza A (H5N1) Vaccine Administered 3 vs. 8 Weeks Apart - A Multi-Center Non-Inferiority Placebo-Controlled Observer-Blinded Phase 2 Randomized Controlled Trial
Brief Title: Immunogenicity and Safety of 2 Doses of Avian Influenza A (H5N1) Vaccine Administered 3 vs. 8 Weeks Apart
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Collaborators: Dalhousie University (Other); IWK Health Centre (Other); Public Health Agency of Canada (PHAC) (Other Government); Canadian Center for Vaccinology (Other); CHU de Quebec-Universite Laval (Other); Vaccine Evaluation Center, Canada (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Joanne Langley, Principal Investigator, Canadian Immunization Research Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT27
Record Dates: First submitted 2025-11-16; First posted 2025-12-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: H5N1 Influenza; H5N1 Virus; Avian Influenza; Avian Influenza A Virus
Keywords: clinical trial; avian flu; H5N1; vaccine
MeSH Terms: conditions — Influenza in Birds | interventions — arepanrix; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: H5N1 vaccines administered 3 weeks apart (Active Comparator): Two doses of the H5N1 vaccine administered 3 weeks apart.
  Normal saline will be administered as a placebo at week 8.
  Interventions: Biological: H5N1 vaccine (Arepanrix); Other: Saline (as a placebo)
- Group 2: H5N1 vaccines administered 8 weeks apart (Active Comparator): Two doses of the H5N1 vaccine administered 8 weeks apart
  Normal saline will be administered as a placebo at week 3.
  Interventions: Biological: H5N1 vaccine (Arepanrix); Other: Saline (as a placebo)

INTERVENTIONS:
Biological: H5N1 vaccine (Arepanrix) — The H5N1 (Arepanrix) vaccine will be administered according to the Product Monograph.
  Other Names: Arepanrix; GSK
Other: Saline (as a placebo) — Normal saline will be administered as a placebo according to the Product Monograph.
  Other Names: Normal Saline

SUMMARY:
Given the recent circulation of avian influenza A(H5N1) clade 2.3.4.4b strains in birds and mammals in North America, Canada procured a supply of Arepanrix™ H5N1 for potential use in persons at high risk of highly pathogenic avian influenza exposure.

This vaccine received regulatory approval in 2013, to be given in two doses at least 3 weeks apart. There is limited data on the effect of various intervals between the two doses on immunogenicity and tolerability. In this study two intervals between doses will be compared (3 vs. 8 weeks apart).

ELIGIBILITY:
Inclusion Criteria:

1. Individuals in stable health (defined as no new onset or exacerbation of pre-existing chronic disease three months prior to vaccination) 18-59 years of age.
2. Able to comply with the trial procedures.
3. Informed consent signed prior to trial-specific procedures.
4. If a person is at risk of becoming pregnant, has practiced adequate contraception for 28 days prior to visit 1, and has a negative pregnancy test on the day of vaccination and has agreed to continue adequate contraception until 60 days after the final vaccination.

Risk of pregnancy is defined as any cis woman and/or gender divergent individual assigned female at birth or with reproductive capacity who is sexually active with individuals with sperm-producing capabilities.

Individual who are post-menopausal or permanently sterile (hysterectomy, bilateral salpingectomy) are not considered at risk of pregnancy. A post-menopausal state is defined as a no menses for 12 months.

Effective contraception methods are:

* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

  * Oral
  * Intravaginal
  * Transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation:

  * Oral
  * Injectable
  * Implantable
* Intra-uterine device (IUD) with or without hormonal release.
* Vasectomised partner, provided that this partner is your sole sexual partner and that the vasectomised partner has received a medical assessment of the surgical success.
* Credible self-reported history of heterosexual abstinence prior to and for at least 28 days after the vaccine.

Effective contraception methods are:

* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

  * Oral
  * Intravaginal
  * Transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation:

  * Oral
  * Injectable
  * Implantable
* Intra-uterine device (IUD) with or without hormonal release.
* Vasectomised partner, provided that this partner is your sole sexual partner and that the vasectomised partner has received a medical assessment of the surgical success.
* Credible self-reported history of heterosexual abstinence prior to and for at least 28 days after the vaccine.

Exclusion Criteria:

* Any of the following:

  1. Receipt of avian influenza A(H5N1) vaccine anytime.
  2. Positive pregnancy test prior to vaccination, or breastfeeding.
  3. Receipt of immunoglobulins and/or any blood products within 3 months preceding the first dose of study vaccine and for one month after the last dose of study vaccine (except Rho D).
  4. Bleeding disorder or history of significant bleeding following IM injections or venipuncture.
  5. Any confirmed or suspected immunosuppressive or immunodeficient state; asplenia, or immunosuppressant medication within the past 6 months except short term oral steroids (≤14 days duration) or topical steroids.
  6. A significant acute disease or temperature ≥38 Co within 24 hours prior to vaccination (temporary exclusion criteria, participants can return for evaluation to be randomized/ vaccinated 72 hours after symptoms resolve).
  7. Unstable chronic medical condition requiring ongoing follow-up and monitoring by a physician as determined by the investigator.
  8. History of anaphylaxis or allergy to any of the constituents or trace residues of the study vaccine, including egg protein.
  9. Receipt of non-study vaccine(s) 2 weeks prior to the study vaccine or planned 2 weeks after administration of the study vaccine.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentages of participants with seroprotection against the H5N1 2.3.4.4b clade vaccine given 3 vs. 8 weeks apart | 28 days post-administration of 2 doses of avian influenza A (H5N1 (Approximately week 12).
  Percentages of participants with seroprotection against the H5N1 2.3.4.4b clade 28 days following administration of 2 doses of avian influenza A(H5N1) vaccine given 3 vs. 8 weeks apart based on serologic outcomes at visit 4 (approximately week 12).
  Seroprotection is defined as the proportion of subjects who were either seronegative prior to vaccination and have a protective post-vaccination HI titre of ≥ 1:40 or who were seropositive prior to vaccination and have at least a 4-fold increase in HI titre post-vaccination.

SECONDARY OUTCOMES:
Immunogenicity - Percentages of participants with seroconversion and the geometric mean fold rise against the H5N1 2.3.4.4b clade vaccine given 3 vs. 8 weeks apart. | 28 days post-administration of 2 doses of avian influenza A (H5N1)
  Definition of Seroconversion rate: the proportion of subjects who were either seronegative prior to vaccination and have a protective post-vaccination HI titre of ≥ 1:40 or who were seropositive prior to vaccination and have at least a 4-fold increase in HI titre post-vaccination) as acceptable by regulators for approval of a Pandemic influenza Vaccine (22).
  Definition of Geometric mean fold rise: the ratio of the post-vaccination geometric mean HI titre divided by the pre-vaccination geometric mean HI titre) acceptable by regulators for approval of a Pandemic influenza Vaccine (22).
Immunogenicity - GMT of HI against the H5N1 2.3.4.4b clade vaccine given 3 vs. 8 weeks apart. | 28 days post-administration of 2 doses of avian influenza A (H5N1) vaccine
  GMT of HI against the H5N1 2.3.4.4b clade 28 days following administration of 2 doses of avian influenza A(H5N1) vaccine given 3 vs. 8 weeks apart.
Immunogenicity - Percentages of participants with seroprotection, seroconversion and the geometric mean fold rise against the H5N1 2.3.4.4b clade | at baseline, at 3 weeks, at 8 weeks, 12 weeks, 26 weeks and through study completion (average of 1 year).
  Percentages of participants with seroprotection, seroconversion and the geometric mean fold rise against the H5N1 2.3.4.4b clade following administration of 1 dose of avian influenza A(H5N1) vaccine.
Immunogenicity - Percentages of participants with seroprotection, seroconversion and the geometric mean fold rise against the H5N1 2.3.4.4b clade | 6 and 12 months after the first dose of avian influenza A (H5N1) vaccine
  Percentages of participants with seroprotection, seroconversion and the geometric mean fold rise against the H5N1 2.3.4.4b clade 6 and 12 months after the first dose of avian influenza A(H5N1) vaccine given 3 vs. 8 weeks apart.
Incidence of Grade 3 & 4 Adverse Events | Up to 12 months after the first dose of avian influenza A (H5N1) vaccine
  The following AEFIs will be collected in all participants:
  1. Grade 3 solicited local and systemic adverse events in the 7 days following vaccine receipt;
  2. SAEs at any time after vaccine receipt during the study;
  3. MAAE at any time after vaccine receipt during the study,
  4. AESI at any time after vaccine receipt during the study;
  5. Provincially reportable AEFI at after vaccine receipt; and
  6. acceptability as measured by participant questionnaire.
  Solicited adverse events and grading Grade 3 and 4 solicited local (injection-site) and systemic adverse events occurring during the 7-day follow-up period after each injection will be recorded.
  Solicited local (injection-site) adverse events (Pain, redness and swelling at injection site).
  Solicited systemic AEs, grade 3 and 4 will be recorded (Fatigue, fever - recorded, headache, nausea, diarrhea, vomiting, generalized muscle aches, joint pain and chills).

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Langley, Principal Investigator — CIRN, Canadian Center for Vaccinology, Dalhousie University
Locations (4):
- Canada (4):
  - Vaccine Evaluation Center, Vancouver, British Columbia
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Vaccine Study Centre of the McGill University Health Centre, Pierrefonds, Quebec
  - CHU de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website with information about study recruitment — https://centerforvaccinology.ca/participate/studies